CLINICAL TRIAL: NCT05549271
Title: Evaluation of the Long-term Efficacy and Safety of the Omega Loop Bypass Versus the Roux-en-Y Gastric Bypass on the Cohort of Patients Included in the Randomized Trial YOMEGA (DGOS 13-0037)
Brief Title: 5 and 7-year Follow-up of the YOMEGA Trial Cohort
Acronym: YOMEGA 5-7y
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 773
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Obesity
Keywords: bariatric surgery; Randomized trial; Roux-en-Y gastric Bypass; One Anastomosis gastric Bypass; long-term results
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obese patients who underwent a Laparoscopic One Anastomosis Gastric Bypass (OAGB) 5 years ago: Patients (BMI > or = 35kg/m2 +/- co-morbidities) who have been operated on using the Gastric bypass procedure built with an Omega loop of 200 cm and a unique gastro-jejunal anastomosis
  Interventions: Procedure: Laparoscopic Mini-gastric bypass
- Obese patients who underwent a Laparoscopic Roux-en-Y Gastric ByPass (RYGBP) 5 years ago: Patients (BMI > or = 35kg/m2 +/- co-morbidities) who have been operated on using the Roux-en-Y gastric bypass which consists in a small gastric pouch (30cc), a 150cm alimentary limb and a 50cm biliary limb. Mesenteric defects were closed.
  Interventions: Procedure: Laparoscopic Roux-en-Y Gastric ByPass (RYGBP)

INTERVENTIONS:
Procedure: Laparoscopic Mini-gastric bypass — The laparoscopic Omega Loop Bypass performed 5 years ago consisted of a long gastric tube, stapled approximately 1.5 cm from the left of the lesser curvature of the antrum to the angle of His, a narrow gastric tube calibrated to be approximately 1.5 cm wide, an Omega loop of 200 cm, a unique gastro-jejunal anatomosis of 200cm from the ligament of Treitz, using a linear stapler
  Groups: Obese patients who underwent a Laparoscopic One Anastomosis Gastric Bypass (OAGB) 5 years ago
Procedure: Laparoscopic Roux-en-Y Gastric ByPass (RYGBP) — The laparoscopic Roux-en-Y Gastric Bypass performed 5 years ago consisted of : a small gastric pouch (about 30cc), an antecolic alimentary limb, a gastro-jejunal anastomosis using a linear stapler, a 150cm long alimentary limb, a 50cm biliary limb, a latero-lateral jejuno-jejunal anastomosis, closure of the mesenteric defects.
  Groups: Obese patients who underwent a Laparoscopic Roux-en-Y Gastric ByPass (RYGBP) 5 years ago

SUMMARY:
Over the last 40 years, the Roux-en-Y Gastric Bypass (RYGB) has been the gold standard in the surgical management of morbid obesity. and is a validated bariatric procedure in France. Nevertheless, the RYGB remains a technically demanding procedure; thus and in order to overcome the complexity of this intervention, a simpler technique based on a single anastomosis at 200cm from the Treitz angle creating an omega loop (Mini Gastric Bypass - MGB or One Anastomosis Gastric Bypass-OAGB) has gradually spread around the worl without prior evaluation, . In 2018, the MGB was officially recognized by the International Federation of Bariatric Surgery (IFSO) as a standard procedure but not by the ASMBS American Society for Metabolic and Bariatric Surgery ; indeed, the OAGB remains controversial because considered by many surgeons at risk of biliary reflux and malnutrition.

DETAILED DESCRIPTION:
Over the last 40 years, the Roux-en-Y Gastric Bypass (RYGB) has been the gold standard in the surgical management of morbid obesity. and is a validated bariatric procedure in France. Nevertheless, the RYGB remains a technically demanding procedure; thus and in order to overcome the complexity of this intervention, a simpler technique based on a single anastomosis at 200cm from the Treitz angle creating an omega loop (Mini Gastric Bypass - MGB or One Anastomosis Gastric Bypass-OAGB) has gradually spread around the worl without prior evaluation, . In 2018, the MGB was officially recognized by the International Federation of Bariatric Surgery (IFSO) as a standard procedure but not by the ASMBS; indeed, the OAGB remains controversial because considered by many surgeons at risk of biliary reflux and malnutrition.

In France, the national and multicenter randomized trial YOMEGA(NCT02139813), comparing the MGB to the RYGB in a prospective randomized fashion confirmed the non-inferiority of MGB compared to the RYGB in terms of weight loss at 24 months. However, significantly more complications (notably at the nutritional level) were observed in the MGB arm.After the publication of these results in September 2019, the High Authority for health (HAS) in France considered that the MGB 200cm did not constitute a validated technique nor an alternative to the RYGB, due to the worrying safety signals. Reimbursement of the MGB was also put into question by the national insurance health care system.

Nevertheless, the use and advantages of the MGB remain a hot topic with several retrospective data showing that a shorter biliopancreatic loop (150cm) would present a lower nutritional risk and excellent weight and metabolic results. A randomized trial comparing the MGB 150cm to the RYGB will thus begin soon in France (YOMEGA-2). The HAS recommends evaluating its efficacy in terms of long-term weight loss, the resolution of comorbidities but also safety outcomes. Finally, patients who have already been operated by MGB must benefit from follow-up with particular vigilance in the detection of nutritional complications and cancer of the lower esophagus. MGB could also turn out to be less expensive than RYGB: shorter operating time and better control of metabolic diseases The scientific community are still awaiting long-term data to reconsider the place of the MGB in the surgical management of obese patients. The aim of our study is to provide long-term efficacy and safety data on the YOMEGA cohort comparing the MGB to the RYGB, at 5 and 7 years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

Patients included in the YOMEGA study, randomized and operated on with the technique assigned to them (121 RYGB and 127 MGB).

The main inclusion criteria for the YOMEGA study were:

* Aged between 18 and 65 years old
* Morbid obesity with BMI ≥ 40 kg/m2 or BMI ≥ 35 kg/m2 associated with one or more co-morbidities (type 2 diabetes, arterial hypertension, sleep apnea, dyslipidemia, arthritis)
* Patient who has benefited from an upper GI endoscopy with biopsies
* Patient who has benefited from a pluridisciplinary evaluation, with a favorable opinion for a gastric bypass
* Patient who understands and accepts the need for a long term follow-up
* Patient who agrees to be included in the study and who signs the informed consent form
* Patient affiliated to a healthcare insurance plan

Exclusion Criteria:

Patients randomized in the YOMEGA study, not operated on with the technique assigned to them.

Main non-inclusion criteria for the YOMEGA study:

* History of esophagitis on upper GI endoscopy (Los Angeles classification)
* Severe gastroesophageal reflux disease (GERD), resistant to medical treatment
* Presence of dysplastic modifications of the gastric mucosa or a history of gastric cancer, on upper gastrointestinal endoscopy.
* Presence of Helicobacter Pylori resistant to medical treatment
* Presence of an unhealed gastro-duodenal ulcer or an ulcer diagnosed less than 2 months previously
* History of previous bariatric surgery (gastric band, sleeve gastrectomy, vertical banded gastroplasty)
* Presence of a severe and evolutive life threatening pathology, unrelated to obesity
* Presence of chronic diarrhea (≥3 loose or liquid stools per day, over a period of more than 4 weeks)
* Pregnancy or desire to be pregnant during the study
* Binge eating disorders or other eating disorders according to DSM V criteria (Diagnostic and Statistical Manual of Mental Disorders)
* Mentally unbalanced patients, under supervision or guardianship
* Patient who does not understand French/is unable to give consent
* Patient not affiliated to a French or European healthcare insurance
* Patient who has already been included in a trial which has a conflict of interests with the present study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in the YOMEGA study, randomized and operated on with the technique assigned to them (121 RYGB and 127 OLB)
Sampling Method: Non-Probability Sample
Enrollment: 248 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Weight loss assessment | 5 and 7 years after surgery
  Measured according to :
  Excess BMI Loss percentage (EBL%), calculated using the following formula:
  ((BMI 5 years after surgery - initial BMI) / (initial BMI - Ideal BMI)) X 100.
  And :
  ((BMI 7 years after surgery - initial BMI) / (initial BMI - Ideal BMI)) X 100. Using 25 as ideal BMI

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - Cabinet de chirurgie générale, digestive et de l'obésité - Hôpital Privé Drôme et Ardèche, Guilherand-Granges
  - Service de Chirurgie Générale et Endocrinienne - Hôpital Claude Huriez - CHU de Lille, Lille
  - Service de Chirurgie Digestive Hôpital Edouard Herriot, Lyon
  - Département de Chirurgie Digestive et Hépatobiliaire - Hôpital Pitié Salpétrière, Paris
  - AP-HP Hôpîtal Europeen Georges Pompidou, Paris
  - Service de Chirurgie Digestive, Générale et Cancérologique - HEGP, Paris
  - Service de Chirurgie Générale - Hôpital Privé de la Loire, Saint-Etienne
  - Service de Chirurgie Générale, Digestive et Viscérale - Centre Hospitalier Intercommunal de Poissy / Saint Gerrmain en Laye, Saint-Germain-en-Laye
  - Département de Chirurgie Digestive et Hépatobiliaire - Centre Hospitalier Privé Saint Grégoire, Saint-Grégoire

REFERENCES:
- [Derived] Robert M, Poghosyan T, Maucort-Boulch D, Filippello A, Caiazzo R, Sterkers A, Khamphommala L, Reche F, Malherbe V, Torcivia A, Saber T, Delaunay D, Langlois-Jacques C, Suffisseau A, Bin S, Disse E, Pattou F. Efficacy and safety of one anastomosis gastric bypass versus Roux-en-Y gastric bypass at 5 years (YOMEGA): a prospective, open-label, non-inferiority, randomised extension study. Lancet Diabetes Endocrinol. 2024 Apr;12(4):267-276. doi: 10.1016/S2213-8587(24)00035-4. Epub 2024 Mar 4. PMID 38452784